CLINICAL TRIAL: NCT00004665
Title: Phase II Study of Long-Term Dehydroepiandrosterone for Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11935; NU-552
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: dehydroepiandrosterone

SUMMARY:
OBJECTIVES:

I. Evaluate the long-term safety and tolerance of a synthetic formulation of dehydroepiandrosterone, GL701, in patients with systemic lupus erythematosus who have completed a prior GL701 protocol.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive daily oral dehydroepiandrosterone for 12 months. The dose is adjusted based on disease activity and tolerance of treatment.

Patients are followed every 3 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Systemic lupus erythematosus by American College of Rheumatology criteria Mild to moderate disease characterized as follows: Prednisone dose (or equivalent) 10 to 30 mg/day No daily dose 1 mg/kg or greater No alternate-day regimen Failed prednisone taper in last 12 months and dose stable for at least 6 weeks prior to entry OR No attempt to taper in last 12 months and dose stable for at least 3 months prior to entry Prior completion of dehydroepiandrosterone (DHEA) study required No prior participation in double-blind DHEA study at Stanford University --Prior/Concurrent Therapy-- No concurrent immunosuppressants No concurrent participation in other clinical studies No investigational agents within the longer of 30 days or 10 half-lives of the agent At least 3 months since immunosuppressants, including: Adrenocorticotropin hormone Androgens Cyclophosphamide Azathioprine Intravenous immune globulin At least 1 month since change in dose of nonsteroidal anti-inflammatory drugs or hydroxychloroquine --Patient Characteristics-- Age: 18 and over Sex: Female only Performance status: Not specified Other: No hypersensitivity to DHEA or inactive ingredient in GL701 formulation, i.e., cornstarch, lactose, or magnesium stearate No condition that would prevent adequate compliance with study No history of breast cancer or reproductive tract malignancy Negative pregnancy test required within 2 weeks prior to entry Reliable contraception required of fertile women No estrogen-containing oral contraceptive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1995-06

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Ramsey-Goldman, Study Chair — Northwestern University